CLINICAL TRIAL: NCT00197067
Title: A Bridging Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Candidate Vaccines RTS,S/AS02D (0.5 mL Dose) and RTS,S/AS02A (0.25 mL Dose) Administered According to a 0, 1, 2 Month Vaccination Schedule in Children Aged 3 to 5 Years Living in a Malaria-endemic Region of Mozambique.
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Candidate Vaccines RTS,S/AS02D (0.5 mL Dose) and RTS,S/AS02A (0.25 mL Dose) Administered IM According to a 0, 1, 2 Month Vaccination Schedule in Children Aged 3 to 5 Years Living in a Malaria-endemic Region of Mozambique.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: 257049/034
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine; RTS,S-AS02A vaccine

INTERVENTIONS:
Biological: RTS,S/AS02D and RTS,S/AS02A
  Other Names: RTS; S/AS02D and RTS; S/AS02A

SUMMARY:
GSK Biologicals is developing in partnership with the Malaria Vaccine Initiative at PATH a candidate malaria vaccine RTS,S/AS02 for the routine immunization of infants and children living in malaria endemic areas. The vaccine would offer protection against malaria disease due to the parasite Plasmodium falciparum and also would provide protection against infection with hepatitis B virus. Studies conducted using the formulation RTS,S/AS02A (0.25 ml dose) in children and adults have shown to be safe. Currently all intramuscular vaccines in the EPI schedule are administered at a dose volume of 0.5 ml and in this context, a new variant of RTS,S/AS02D (0.5 ml dose) formulation has been composed which has the same active constituents in the same quantities as in a 0.25 ml dose of RTS,S/AS02A. In this study, RTS,S/AS02D (0.5 ml dose) was compared to the existing formulation, RTS,S/AS02A (0.25 ml dose).

DETAILED DESCRIPTION:
Children participating in this study will either receive RTS,S/AS02D (0.5 ml dose) or RTS,S/AS02A (0.25 ml dose) intramuscularly according to 0, 1, 2 months schedule. The children will be followed-up throughout the study period to record safety events. Blood samples will be collected at defined time points to assess the subject's immune response to the relevant immunological indicators.

ELIGIBILITY:
Inclusion criteria:

Healthy children of both sexes between the ages of 3 to 5 years (up to but not including 6th birthday) who had not previously been immunized with hepatitis B vaccine, whose parents or guardians the investigator believed could and would comply with the requirements of the protocol, whose parents or guardians would give written or oral, signed or thumb printed and witnessed informed consent, who were free of obvious health problems as established by medical history and clinical examination before entering into the study and who were available for the foreseen duration of the immunization and follow-up period.

Exclusion criteria:

If the child was found to have major congenital defects or serious chronic illness; history of surgical splenectomy; a diagnosis or clinical suspicion of an immunosuppressive or immunodeficient condition; family history of congenital or hereditary immunodeficiency; history of allergic disease or reactions likely to be exacerbated by any component of the vaccine; previous vaccination with hepatitis B vaccines or with an experimental vaccine; or if the child is simultaneously participating in any other clinical trial, then the child would be excluded from the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2004-03-15 (Actual); Primary Completion 2005-04-26 (Actual); Study Completion 2005-04-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited symptoms and serious adverse events during the entire study period; to assess antibody levels for relevant immunological indicators at time points when post completion of vaccination schedule.

SECONDARY OUTCOMES:
To assess antibody levels for relevant immunological indicators at time points when blood sampling will be done.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD for this study is available via the Clinical Study Data Request site.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=19808

REFERENCES:
- See also: Results for study 257049/034 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/257049/034?search=study&#rs